CLINICAL TRIAL: NCT03667118
Title: Daily Ingestion of a Multi-Allergen Food Supplement by Infants: Clinical Symptoms, Reactions, and Acceptability - A Randomized Trial
Brief Title: Introduction and Maintenance of Still Eating Protein Blends in Support of Infant Nutritional Goals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jane Holl, Director, Center for Healthcare Studies, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00205862
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant
Masking Description: Parents received packets of the powder to be fed from their infant directly from the manufacturer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Supplement (Experimental): Infants who received the active food supplement powder
  Interventions: Dietary Supplement: Food Supplement
- Placebo (Placebo Comparator): Infants who received the placebo powder
  Interventions: Dietary Supplement: Food Supplement

INTERVENTIONS:
Dietary Supplement: Food Supplement — A powder blend of 16 common allergenic proteins ([oat, milk, egg, sesame, wheat] [almond cashew, hazelnut, peanut, pecan, pistachios, soy, walnut] [cod, shrimp, salmon]) combined with 400 IU of Vitamin D3

SUMMARY:
The purpose of the study is to test a food supplement to:

* Show that the food supplement is well tolerated and safe to feed to infants;
* Find out how often parents/caregivers feed their infants the food supplement;
* Find out how parents/caregivers usually add the food supplement to infants' regular solid or liquid food; and
* Learn what aspects of the food supplement are more or less attractive to infants and to parents/caregivers.

DETAILED DESCRIPTION:
The study involves parents/caregivers of infants, ≥ 5 months but < 11 months of age. Parents who enrolled their infants complete a 1-month blinded placebo run-in period, followed by randomization to placebo or the food supplement.

During the intervention period, infants randomized to the food supplement are fed a once daily, individual packet of the food supplement mixed into liquid (e.g., breast milk, infant formula) or solid (e.g., applesauce, pureed carrots) foods being fed to the infant. The food supplement is a blend of 16 common allergenic proteins ([oat, milk, egg, sesame, wheat] [almond cashew, hazelnut, peanut, pecan, pistachios, soy, walnut] [cod, shrimp, salmon]) combined with 400 IU of Vitamin D3. Parents complete a daily diary about any reactions or symptoms within 2 hours of ingesting the food supplement. Infants randomized to the placebo are also fed a once daily individual packet of the placebo mixed into liquid or solid foods being fed to the infant. Parents also complete a daily diary about any reactions or symptoms within 2 hours of ingesting the placebo.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants, ≥ 5 months but < 11 months of age whose parent/caregiver can provide, in English, consent, understand instructions and complete a daily diet diary for their child, answer questions about how much and in what food they mix the Food supplement, and report any reaction or adverse event. Pregnant women will not be excluded if they have a child who is eligible for the study.

Exclusion Criteria:

* - Any parent/caregiver who cannot provide consent.
* Any parent/caregiver who cannot understand or write English.
* A parent/caregiver who is in prison.
* Any infant who

  * Has a previous or current diagnosis of food allergy, made by a board-certified allergy and immunology specialist;
  * Was born before 37 weeks of pregnancy (premature birth);
  * Has severe eczema, as determined by two parent/caregiver questions:

    1. During the past 6-11months, have you been told by a doctor or other health professional that your infant has eczema or any kind of skin allergy? (National Health Interview Survey, 2012) If yes, go to Question 2.
    2. Would you describe (his/her) eczema or skin allergy as mild, moderate, or severe? (National Survey of Children's Health, 2007) If described as severe, infant is excluded.
  * Has a current serious, chronic condition, as measured by:

    1. Does you infant have a health condition that has lasted for more than three (3) months? If yes, go to Question 2.
    2. Has your infant been hospitalized more than 2 times since birth for this condition? If yes to Question 1 and 2, infant is excluded.
* If a parent/caregiver has multiple birth infants (e.g., twins), only one eligible infant will be selected.
* Any person who works for Before Brands or who has a family member working for Before Brands.

Ages: 5 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 705 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Allergic-type reaction | 1month
  difference between the proportion of infants with allergic-type reaction within 2 hours of ingestion in the food supplement versus placebo arm

SECONDARY OUTCOMES:
Symptom | 1 month
  difference between the proportion of infants with a symptom within 2 hours of ingestion of the food supplement versus placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Jane L Holl, MD MPH, Principal Investigator — Professor of Pediatrics, Feinberg School of Medicine
Locations (1):
- Jane L Holl, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Demographic data about the study participants Outcomes of the study